CLINICAL TRIAL: NCT01050361
Title: Echocardiography-Guided Hemodynamic Management Strategy for Patients Requiring Perioperative Care for Non-Cardiac Surgery
Brief Title: Echocardiography Management for Patients Requiring Care for Non-Cardiac Surgery
Acronym: EGHEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0321-09-FB
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Risk Factors
Keywords: congestive heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Echo Guided HEmodyanmic Management (EGHEM) (Experimental): EGHEM - Echo Guided HEmodyanmic Management - will receive their intraoperative maintenance fluid and possible drug therapy (furosemide) based on their hourly intraoperative Left Ventricular Diastolic Dysfunction (LVDD) grade.
  Interventions: Procedure: Transthoracic Echocardiogram (TTE)/Transesophageal Echocardiogram (TEE)
- Standard HEmodynamic Management (SHEM) (No Intervention): SHEM - Standard HEmodynamic Management - will NOT receive the study intervention, but will receive standard anesthesia and hemodynamic management based on current standards within the institution (control group).

INTERVENTIONS:
Procedure: Transthoracic Echocardiogram (TTE)/Transesophageal Echocardiogram (TEE) — Duration lasts the entire operation.
  Arms: Echo Guided HEmodyanmic Management (EGHEM)

SUMMARY:
The growing population of institution patients with heart failure combined with the increasing number of surgical procedures performed each year supports the need for a critical analysis of how to most appropriately manage these patients during the perioperative period, especially for non-cardiac surgery. Echo-guided hemodynamic management (EGHEM) is the use of echocardiography data to normalize and/or optimize in real-time, cardiac output and ventricular filling pressures in the perioperative period for non-cardiac surgical cases. The purpose of this study is to test the hypothesis that EGHEM compared to standard management practices will result in a reduced length of hospital stay in the noncardiac surgery population. The primary goal of health care providers for patients requiring anesthetic care, perioperative care, or critical care is ensuring the adequacy of the patient's circulatory function by optimizing cardiac output and ventricular filling pressure. Currently, the use of the ECG monitor and systemic blood pressure are the standard of care for assessing circulatory function. However, those data cannot provide accurate information on cardiac output and ventricular filling pressure for patients with cardiovascular risk factors and/or comorbidities. As a result, managing the hemodynamic parameters of these patients, as well as their intravenous fluid needs and resuscitation strategy, we hypothesize that using traditional approaches may lead to significant volume overload and post-operative cardiovascular complications and morbidity. In this study we propose an EGHEM strategy that incorporates standard echocardiography generated data points in addition to the systemic blood pressure and ECG signal to assess, manage, modify and optimize patient cardiac preload, afterload, heart rate and contractility in the perioperative period. Based on our initial observations and preliminary data using the EGHEM approach, we hypothesize that we can demonstrate a significant decrease in hospital length of stay and an overall decrease in perioperative morbidity at 30 days in the non-cardiac surgery population using EGHEM compared to standard practices. In this proposal we have designed a single center, prospective, randomized clinical trial to test our hypothesis.

DETAILED DESCRIPTION:
Step 1: Patient selection

The first step in the EGHEM/EGAM process is appropriate patient selection. Patients who have any of the following cardiovascular risk factors and/or comorbidities and are scheduled for a non-cardiac surgery are candidates for EGHEM/EGAM:

1. Urology/gynecology/General surgical patient
2. Non-cardiac surgical population
3. age 65 years or older, OR 19 years or older and one of the following risk factors:

   1. Hypertension (HTN)
   2. Diabetes
   3. Obesity (body mass index [BMI] >35)
   4. Renal insufficiency
   5. Tobacco usage
   6. Hypercholesterolemia
   7. Sleep apnea/heavy snoring at night
   8. Clinical diagnosis of congestive heart failure (CHF) as defined by:

      * Dyspnea on exertion
      * Paroxysmal nocturnal dyspnea
      * Orthopnea
      * Elevated jugular venous pressure
      * Pulmonary rales
      * Third heart sound
      * Cardiomegaly or pulmonary edema on chest x-ray
      * Peripheral edema
      * Hepatomegaly
      * Pleural effusion
   9. Palpitations/irregular heart beats
   10. Chest pain at rest and or exercise
   11. Murmur on examination
   12. Known coronary artery disease (CAD)/stents/coronary artery bypass graft (CABG)
   13. Known valvular disease
   14. Known stroke or transient ischemic attacks (TIA) Standard Medical Care Step 2: Pre-op assessment

Step 2 in the EGAM process involves a bedside, transthoracic echocardiography (TTE) pre-op assessment. The pre-op TTE should be performed by one of the co-investigators, and take less than 10 minutes to complete. The information acquired by TTE during the pre-op assessment should include the following five evaluations, in order of importance:

1. Cardiac output on the left side of the heart using spectral Doppler measurements;

   1. Left ventricular outflow tract (LVOT) velocity time integral (VTI)
   2. Heart rate
2. Filling pressures on the left side of the heart using spectral Doppler measurements;

   1. The pulmonary venous flow pattern defined as co-dominant, systolic dominant or diastolic dominant
   2. The mitral inflow pattern defined as normal, impaired relaxation, pseudonormal or restrictive
   3. The E/e' ratio of velocities
3. Mitral valve structure and function;
4. Aortic valve structure and function; and
5. Biventricular contractility.

These evaluations are performed using the following TTE views:

A. Parasternal (PS) window: With the patient in the left lateral decubitus position, the TTE probe is placed on the 3rd left intercostal space next to the sternum; the light on the probe should be directed toward the patient's right shoulder. The 2-dimensional image of the long axis (LAX) should be acquired first. In this view, the following are evaluated:

* Color Doppler on aortic valve (AV) and mitral valve (MV)
* E-point septal separation (EPSS) To evaluate the PS short axis (SAX), the probe should be rotated clockwise 60 degrees. The 2-dimensional view should be obtained at the mid-papillary level.

B. Apical window: With the patient in the same left, lateral, decubitus position, the probe is placed between the 5th and 6th intercostal space on the left side, close to the nipple line. The light on the probe should be directed toward the floor or the bed for the 4-chamber view. The following assessments should be performed in the 4-chamber view:

* Two-dimensional image;
* Pulsed-wave (PW) Doppler in the right upper pulmonary vein;
* PW Doppler at the tip of the MV;
* PW Doppler on the MV annulus for tissue Doppler;
* Color Doppler on the tricuspid valve (TV) and MV if necessary based on the PS LAX window.

For the apical LAX, the probe should be rotated counterclockwise so that the light is directed toward the patient's right shoulder. In the LAX view, velocity time integrals (VTIs) using PW in the left ventricular outflow track (LVOT) and continuous wave (CW) at the level of the AV should be acquired.

C. Subcostal window: With the patient supine, the TTE probe is placed under the right costal ridge and directed toward the heart. The light should be directed toward the sonographer (toward the patient's left) to assess the 4-chamber view.

For the subcostal inferior vena cava (IVC) view, the probe should be slightly rotated counterclockwise until the IVC can be assessed.

Standard Medical Care Step 3: Management strategies Step 3 in the EGHEM/EGAM process is to define patient management strategies based on the pre-op TTE assessment. The main goals of patient management are to maintain normal cardiac output and filling pressure. Primary and secondary findings and the associated EGAM strategies to achieve these goals are outlined in Table 1 and Table 2, respectively.

Table 1: Primary findings and associated management strategy to maintain normal cardiac output and filling pressure.

Echo-Generated Findings EGHEM/EGAM Strategy Cardiac output status Filling pressure status Normal High Preload reduction Low Normal Afterload reduction Low High Afterload and preload reduction High High Preload reduction High Normal or low Increase preload

Table 2: Secondary findings and associated management strategy to optimize patient management.

Echo-Generated Finding EGHEM/EGAM Strategy Filling Pressure Other High Aortic stenosis Preload reduction Normal Aortic stenosis Safe for afterload reduction

* Mitral regurgitation Afterload reduction
* Low contractility Inotropic support
* Suspected or confirmed CAD Maintain heart rate in the 50 - 60 bpm range right ventricle (RV) volume overload Preload reduction RV pressure overload Pulmonary afterload reduction Standard Medical Care Step 4: Ongoing intra-operative assessment Based on the appropriate EGAM strategy defined in Step 3, either TEE or TTE should be used during the surgical procedure for the ongoing patient assessment every 15 to 20 minutes. The PI or Secondary Investigator will determine whether a TEE or TTE should be conducted intra-operatively. The results of these tests will be used for research purposes. During surgery: fluid administration, afterload adjustments, and supported contractility can be implemented to optimize patient management. It is difficult to assess cardiac output with the current standard medical care without invasive monitoring. There is minimal risk if the physician gets distracted by the echocardiogram or the algorithm of the study however it is unlikely this tool would be a distraction to the physician as it is monitoring the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years
2. Hypertension (HTN)
3. Diabetes
4. Obesity (body mass index [BMI] >35)
5. Renal insufficiency
6. Tobacco usage
7. Hypercholesterolemia
8. Sleep apnea/heavy snoring at night
9. Clinical diagnosis of CHF as defined by:

   1. Dyspnea on exertion
   2. Paroxysmal nocturnal dyspnea
   3. Orthopnea
   4. Elevated jugular venous pressure
   5. Pulmonary rales
   6. Third heart sound
   7. Cardiomegaly or pulmonary edema on chest x-ray
   8. Peripheral edema
   9. Hepatomegaly
   10. Pleural effusion
10. Palpitations/irregular heart beats
11. Chest pain at rest and or exercise
12. Murmur on examination
13. Known coronary artery disease (CAD)/stents/coronary artery bypass graft (CABG)
14. Known valvular disease
15. Known stroke or transient ischemic attacks (TIA)

Exclusion Criteria:

1. Patients expected to say in the hospital for less than 24 hours.
2. Inability of undergo TEE and TTE
3. Clinical evidence or suspicion of elevated intracranial pressure.
4. Preoperative shock or systemic sepsis
5. Emergency Operation
6. American Society of Anesthesiologists (ASA) Class V
7. Inability of give informed consent
8. Participation in another clinical trial
9. Prisoner

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2013-01-09 (Actual); Study Completion 2013-01-09 (Actual)

PRIMARY OUTCOMES:
Optimizing participant perioperative hemodynamic management (cardiac ultrasound) | 3 Years
  Obtain standard cardiac ultrasound-generated data points [Parasternal Long Axis, Parasternal Short Axis, Apical 4 Chamber, Subxiphoid (Subcostal), and inferior vena cava (IVC) views] to manage, modify, and optimize the participant cardiac preload, afterload, heart rate and contractility in the perioperative period.
Perioperative morbidity in congestive heart failure for non-cardiac surgeries | 3 years
  Incidence of perioperative morbidity associated with congestive heart failure for non-cardiac surgeries.
Evaluate echocardiography technology for identifying participant perioperative hemodynamic management needs | 3 years
  To evaluate and support the conclusion that echocardiography is a superior technology for identifying these changes and managing the unique cardiovascular challenges of the patient population.
Reducing perioperative mortality in congestive heart failure for non-cardiac surgeries | 3 years
  Perioperative mortality associated with congestive heart failure for non-cardiac surgeries.
Optimizing participant perioperative hemodynamic management (systemic blood pressure) | 3 Years
  Obtain standard systemic blood pressure (normal: systolic pressure of less than 120 and a diastolic pressure of less than 80, elevated: systolic pressure between 120 and 129 with a diastolic pressure of less than 80) to manage, modify, and optimize the participant cardiac preload, afterload, heart rate and contractility in the perioperative period.
Optimizing participant perioperative hemodynamic management electrocardiogram (ECG signal) | 3 Years
  Obtain standard electrocardiogram (ECG: normal values defined as follows: P-wave axis 0° to 75°, QRS axis -30° to 90°, and T axis 15° to 75) to manage, modify, and optimize the participant cardiac preload, afterload, heart rate and contractility in the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Tara R Brakke, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States